CLINICAL TRIAL: NCT03154983
Title: The Clinical Research of Mesylate Apatinib Combined With Docetaxel and S-1 as the First-line Treatment of Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhou Fuxiang (Other)
Collaborators: Hubei Cancer Hospital (Other); Huangshi Central Hospital (Other); The Central Hospital of Huanggang (Other); Xianning Central Hospital (Other); Taihe Hospital (Other); The first hospital of Zaoyang (Unknown); Hanchuan City people's Hospital (Unknown); Yangxin People's Hospital (Unknown); Tianmen People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Zhou Fuxiang, Director, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC G04
Record Dates: First submitted 2017-05-08; First posted 2017-05-16 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Gastric Cancer
Keywords: Mesylate Apatinib; The First-line Treatment; Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Tegafur; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-line treatment (Experimental): First-line treatment：treatment including Mesylate Apatinib Combined With Docetaxel and S-1(DS).DS Docetaxel 75mg/m2 d1 iv.drop 1h（one hour）， S-1(BSA<1.25 40mg Po bid(twice a day), BSA >=1.25-<1.5 50mg Po bid, BSA >=1.5 60mg Po bid), Q21d(21 days a cycle); Mesylate Apatinib 500mg Po QD(once a day) continuous use; until disease deterioration.
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel — Diagnosed with metastatic gastric cancer patients (including the esophagogastric junction adenocarcinoma), DS(docetaxel and Tegafur)and Mesylate apatinib 6 cycles, the specific amount of usage: DS Docetaxel 75mg/m2 D1 IV.drop 1H（one hour）, Tegafur(BSA<1.25 40mg Po bid(twice a day), BSA >=1.25-<1.5 50mg Po bid, BSA >=1.5 60mg Po bid, Q21d(21 days a cycle)); Mesylate Apatinib 500mg Po QD（once a day)） continuous use, until disease deterioration.
  Other Names: Tegafur; Mesylate Apatinib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Apatinib Mesylate Tablets combined with docetaxel and S-1 as the first-line treatment of metastatic gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years of age;
2. recurrent or metastatic adenocarcinoma of the stomach or gastroesophageal junction diagnosed by pathology (including histology or cytology);
3. 1 measurable lesions at least should be detected by CT/MRI examination in accordance with the RECIST(Response Evaluation Criteria In Solid Tumors）1.1;
4. had not received other anti VEGFR targeted therapy;
5. ECOG（Eastern Cooperative Oncology Group）PS（Performance Status）:0-2 scores;
6. the expected survival time is more than 3 months;
7. if patient had accepted the chemotherapy, the time from the last chemotherapy should be more than 6 months;
8. the damage caused by other treatments has been restored, and the subjects received radiotherapy or surgery over 4 weeks ago, and the wound has healed completely;
9. the main organ function is normal, which should meet the following criteria: (1) blood routine examination standards should be met: (no blood transfusion within 14 days) A. HB（hemoglobin） = 90g/L, B. ANC(absolute neutrophil count) = 1.5 * 109/L, C. PLT（platelet） = 80 * 109/L; (2) biochemical examination shall comply with the following criteria: A. BIL（bilirubin） <1.25 normal upper limit (ULN), B. ALT（glutamic-pyruvic transaminase） and AST（glutamic-oxalacetic transaminase）<2.5ULN（upper limit of normal）, if subjects have liver metastases, the ALT and AST <5ULN（upper limit of normal）, C. Cr ≤ 1ULN, CCR（creatinine clearance rate） > 50ml/min (Cockcroft-Gault formula);
10. women of childbearing age must have a pregnancy test in 7 days before entering the group (in serum), and the results were negative, and willing to use appropriate contraception during the study period and the last 8 weeks after giving drug test; men should have the surgical sterilization, or adopt the appropriate contraceptive methods during the test and the last 8 weeks after giving drug test;
11. participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up.

Exclusion Criteria:

1. Suffering from other malignant tumors previously or at the same time, with the exception of cured skin basal cell carcinoma and cervical carcinoma in situ;
2. Patients have used the paclitaxel class and / or S-1 as the adjuvant therapy in 2;
3. have been confirmed to be allergic to docetaxel, 5-fluorouracil, apatinib and / or its accessories;
4. the blood pressure of patients with hypertension cannot be reduced to the normal range by the antihypertensive drugs (systolic pressure >140 mmHg, diastolic pressure >90 mmHg);
5. patients are suffering from severe cardiovascular disease: the II level of myocardial ischemia or myocardial infarction, poor control of the arrhythmia (including QTc(corrected QT interval) prolongation of male > 450 ms, of female > 470ms ); and patients have III-IV grade of cardiac insufficiency, or left ventricular (LVEF) < 50% shown by echocardiography according to the NYHA(New York Heart Association) standard;
6. patients are positive of urine protein (urine protein detection 2+ or above, or 24 hours urine protein quantitative >1.0g);
7. have a variety of factors that affect oral drugs (such as difficulty in swallowing, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.);
8. patients have a clear tendency with gastrointestinal bleeding, including the following situation: local active ulcerative lesions, and fecal occult blood (+ +); with melena and hematemesis history in 2 months; and patients with fecal occult blood (+) and unresected gastric primary tumor; patients with the risk of bleeding should take the gastroscopy test, if it is the gastric cancer, and researchers believe that may results in massive digestive tract hemorrhage;
9. coagulation dysfunction (INR(international normalized ratio)>1.5, APTT(activated partial thromboplastin time)>1.5 ULN), with bleeding tendency;
10. patients with a history of psychotropic substance abuse and unable to give up or have mental disorders;
11. Patients who participated in other clinical trials within 4 weeks;
12. have received the VEGFR inhibitors, such as sorafenib and sunitinib;
13. according to the researcher's judgment, there are other accompanying disease endangering the patient's safety or affect the patient to complete the study.
14. patients with central nervous system metastasis;
15. pregnant or lactating women;
16. the researchers consider those who were not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
progress-free survival time | 30 months
  During the treatment, the investigators will arrange patients to underwent CT and MRI examination on time, evaluating the size and the number of the tumor, to determine whether the disease progress than before; and the time from the start of treatment to the progression is progress-free survival time.

SECONDARY OUTCOMES:
Overall survival Time | 30 months
  During and after treatment, all patients were followed up regularly ,the patients will be arranged to evaluate the Performance status score or Karnofsky Performance Score to assess the patient's health and disease controling, until the patient died; the time from the beginning of treatment to death is overall survival time.
Overall remission Rate | during 6 cycles of chemotherapy (each cycle is 28 days)
  During the treatment, the investigators will regularly arrange patients to underwent CT, MRI ,Tumor marker examination and so on, evaluating the size and the number of the tumor, utilizing Response Evaluation Criteria in Solid Tumors to assess whether the disease progress than previous; and the percentage of patients with complete remission and partial remission of the disease is Overall remission Rate.
adverse events | up to 28 weeks
  During and after treatment, the investigators will on the basis of The clinical application expert consensus of Mesylate Apatinib to cure gastric cancer and The evaluation criteria of adverse drug reaction to assess patients who accepted treatment whether has adverse events.
Quality of life | 30 months
  During and after treatment, the investigators will on the basis of The Lancashire Quality of Life Profile to assess the patients' life quality regularly.
disease control rate | 30 months
  During the treatment, the investigators will regularly arrange patients to underwent CT, MRI ,Tumor marker examination and so on, to assess the size and the number of the tumor, utilizing Response Evaluation Criteria in Solid Tumors to assess whether the disease progress than previous; and the percentage of patients with disease control is disease control rate.

CONTACTS AND LOCATIONS:
Overall Officials: Fuxiang Zhou, M.D., Study Chair — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No